CLINICAL TRIAL: NCT04690855
Title: A Multi-institutional Phase II Study to Evaluate Efficacy and Safety of TAlazoparib, Radiotherapy and Atezolizumab in gBRCA 1/2 Negative Patients With PD-L1+ Metastatic Triple Negative Breast Cancer
Brief Title: A Study to Evaluate TAlazoparib, Radiotherapy and Atezolizumab in gBRCA 1/2 Negative Patients With PD-L1+ Metastatic Triple Negative Breast Cancer
Acronym: TARA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study has been terminated due to Lack of Accrual.
Sponsor: Mylin A. Torres, MD (Other)
Collaborators: Genentech, Inc. (Industry); Pfizer (Industry); Emory University (Other)
Responsible Party: Sponsor-Investigator, Mylin A. Torres, MD, Sponsor-Investigator, Hoosier Cancer Research Network
Organization: Hoosier Cancer Research Network (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCRN BRE19-433
Record Dates: First submitted 2020-12-28; First posted 2020-12-31 (Actual); Results first posted 2023-12-04 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Breast Cancer; Triple Negative Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — talazoparib; atezolizumab; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Study Treatment Arm (Experimental): All patients will be treated with induction talazoparib of 1mg PO daily starting Day 1. Patients will then receive 8 Gy x 3 fractions to 1-4 metastatic lesions beginning Day 12,13, or 14 and given QOD. 840 mg of atezolizumab will be given intravenously (IV) on Day 15 of the 1st cycle and then on Day 1 and Day 15 of the remaining cycles. The sequence of administration is not specified on the days in which talazoparib and atezolizumab are given on the same day. Each cycle equals 28 days. Treatment will continue until progression or severe toxicity.
  A safety lead in of up to 6 patients will be performed. Immune-related and non-immune related adverse events will be tracked up to 12 weeks post initiation of atezolizumab, as the majority of treatment-related toxicities from talazoparib, radiation, and atezolizumab occur within this time period.
  Interventions: Drug: Talazoparib; Drug: Atezolizumab; Radiation: Radiation

INTERVENTIONS:
Drug: Talazoparib — Talazoparib 1 mg Orally Day 1 to Day 28
  Other Names: Talzenna
Drug: Atezolizumab — Atezolizumab 840 mg IV over 60 minutes Day 15 of Cycle 1 then Day 1 and Day 15 of subsequent Cycles
  Other Names: Tecentriq
Radiation: Radiation — Radiation 8 Gy will be given in 3 fractions QOD beginning Day 12, 13 or 14 of Cycle 1 but 24-72 hours prior to 1st dose of Atezolizumab

SUMMARY:
This is a Phase II study designed to assess efficacy and safety of talazoparib, high dose radiation, and atezolizumab in patients with metastatic TNBC that is PD-L1 positive. A total of 23 gBRCA pathogenic variant negative patients will be enrolled. All patients will be treated with induction talazoparib of 1mg PO daily starting Day 1. Patients will then receive 8 Gy x 3 fractions to 2-4 metastatic lesions beginning Day 12,13, or 14 and given QOD. 840 mg of atezolizumab will be given intravenously (IV) on Day 15 of the 1st cycle and then on Day 1 and Day 15 of the remaining cycles. The sequence of administration is not specified on the days in which talazoparib and atezolizumab are given on the same day. Each cycle equals 28 days. Treatment will continue until progression or severe toxicity.

A safety lead in of up to 6 patients will be performed. Immune-related and non-immune related adverse events will be tracked up to 12 weeks post initiation of atezolizumab, as the majority of treatment-related toxicities from talazoparib, radiation, and atezolizumab occur within this time period.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide written informed consent/assent and HIPPA for the trial.
2. Ages 18-75 years old at time of consent. Female or male patients allowed.
3. ECOG PS of 0-2, KPS >/= 60%.
4. Biopsy proven metastatic triple negative breast cancer (estrogen receptor (</=10%), progesterone receptor (</=10%) and no overexpression of HER2 as evaluated by local institutions with at least 2 exracranial lesions of metastatic disease on imaging.
5. PD-L1 positive tumor infiltrate as defined as >/= 1% on IHC using the SP142 Ventana Assay.
6. Known gBRCA 1/2 status (gBRCA 1/2 negative [e.g. gBRCA wild-type, gBRCA variants of uncertain significance] are eligible).
7. Patients must have at least 1 extracranial metastatic lesion (may be measurable or non-measurable disease by RECIST v 1.1) that is amenable to high dose radiotherapy and at least one additional extracranial lesion of measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST v1.1) that will not receive radiotherapy on this study. Of note, lesions maybe in the same organ but must be 2 cm apart and breast lesions may be treated.
8. Patients must have received at least one and no more than three previous lines of systemic treatment in the advanced setting with or without immune therapy. Patients with disease recurrence or progression following neoadjuvant or adjuvant cytotoxic chemotherapy are not eligible unless they have received at least one line of chemotherapy with or without immune therapy in the advanced setting. NOTE: Targeted small molecules (e.g. tyrosine kinase inhibitors), hormonal agents and monoclonal antibodies that inhibit angiogenesis (e.g. bevacizumab, afilbercept) are not counted in the number of lines of therapy. Cytotoxic chemotherapy with or without immune therapy for advanced disease prior to protocol treatment is not permitted within 2 weeks of the protocol treatment. Patients may or may not have received radiotherapy or neoadjuvant or adjuvant chemotherapy in the treatment of their initial, non-metastatic breast cancer, but must be entered on study 2 weeks after their last dose of radiotherapy, last cycle of chemotherapy and biologic therapy (if applicable) for mTNBC and have sufficient resolution of side effects per physician assessment at time of talazoparib.
9. Demonstrate adequate organ function as defined in the table below. All screening labs to be obtained within 14 days prior to registration.

   * Absolute neutrophil count > 1500/mcL
   * Platelets >/= 100,000 mm
   * Anemia >/= 9.0 g/dL (NOTE: The use of transfusion or other intervention to achieve Hgb >/= 9.0g/dl is acceptable)
   * Serum creatinine ≤ 1.5 × upper limit of normal (ULN) or calculated creatinine clearance ≥ 60 mL/min using Cockcroft-Gault equation for patients with creatinine levels > 1.5× institutional ULN
   * Total bilirubin ≤ 1.5× ULN OR direct bilirubin ≤ 1× ULN
   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5× ULN unless liver metastases are present, in which case they must be ≤ 5×ULN
   * International normalized ratio (INR) or prothrombin time (PT) ≤1.5× ULN unless patient is receiving anticoagulant therapy as long as PT or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants
   * Activated partial thromboplastin time (aPTT) ≤ 1.5× ULN unless patient is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
10. Patients must be eligible for radiotherapy, talazoparib, and atezolizumab.
11. Females of childbearing potential must have a negative serum or urine pregnancy test within 14 days prior to Cycle 1 Day 1. If a urine test is done and it is positive or cannot be confirmed as negative, a serum pregnancy test will be required. NOTE: Females are considered of child bearing potential unless they are surgically sterile (have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are naturally postmenopausal for at least 12 consecutive months.
12. Women of childbearing potential and males must agree to use two effective methods of contraception or complete abstinence, from the time of signing the informed consent (females) or first day of study treatment (males), during the course of the study and for 7 months (females) and for 4 months (males) after the last dose of study drug.
13. Patients must not have active wound healing issues from surgery and sufficient resolution of surgical side effects, per physician assessment, at time of radiotherapy.
14. During participation on this study, no other investigation or commercial agents or therapy for cancer other than bisphosphonate, rank ligand inhibitors, atezolizumab, radiotherapy and talazoparib should be administered. NOTE: Patients may have received bisphosphonates or rank ligand inhibitors prior to and while on enrollment on study.
15. Patients must have the psychological ability and general health that permits completion of the study requirements and required follow up.

Exclusion Criteria

1. gBRCA1/2 pathogenic variant positive
2. Four or more lines of cytotoxic chemotherapy for mTNBC.
3. Previous radiation to the metastases to be treated with radiation on this protocol.
4. Previous PARPi treatment (e.g. talazoparib, niraparib, olazaparib).
5. Progression of breast cancer within the first 3 months of prior immune therapy for non-metastatic or metastatic breast cancer.
6. Untreated CNS disease (patients with stable CNS disease for at least 28 days and asymptomatic treated CNS metastases are permitted).
7. History of leptomeningeal disease.
8. History of autoimmune disease that has required systemic treatment (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
9. Use of systemic glucocorticoid or immunosuppressive medications at time of enrollment.
10. Severe, active co-morbidity such as CHF or unstable angina within last 6 months, transmural MI within the last 6 months.
11. Acute bacterial or fungal infection requiring IV antibiotics at time of registration.
12. COPD or other respiratory illness requiring hospitalization at time of registration.
13. HIV positive with CD4 count <200 cells/ microliter.
14. Current hormone replacement therapy use.
15. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy. Indolent cancers (such as low risk prostate or in-situ cancers) that are not being treated, are acceptable.
16. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
17. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
18. Receipt of the last dose or treatment of anti-cancer chemotherapy, radiotherapy, surgery, endocrine therapy, targeted therapy, biologic therapy, or tumor embolization ≤ 2 weeks (4 weeks for any monoclonal Antibody (mAb), 6 weeks for nitrosoureas or mitomycin C) prior to first dose of study treatment, or has not recovered (i.e., to ≤Grade 1 or Baseline) from clinically significant adverse events (AEs) due to these previously administered agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2021-10-04 (Actual); Primary Completion 2022-02-18 (Actual); Study Completion 2022-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mylin Torres, MD, Principal Investigator — Winship Cancer Institute, Emory University
Locations (2):
- United States (2):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Winship Cancer Institute of Emory University, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Treatment Arm: All patients will be treated with induction talazoparib of 1mg PO daily starting Day 1. Patients will then receive 8 Gy x 3 fractions to 1-4 metastatic lesions beginning Day 12,13, or 14 and given QOD. 840 mg of atezolizumab will be given intravenously (IV) on Day 15 of the 1st cycle and then on Day 1 and Day 15 of the remaining cycles. The sequence of administration is not specified on the days in which talazoparib and atezolizumab are given on the same day. Each cycle equals 28 days. Treatment will continue until progression or severe toxicity.
  A safety lead in of up to 6 patients will be performed. Immune-related and non-immune related adverse events will be tracked up to 12 weeks post initiation of atezolizumab, as the majority of treatment-related toxicities from talazoparib, radiation, and atezolizumab occur within this time period.
  Talazoparib: Talazoparib 1 mg Orally Day 1 to Day 28
  Atezolizumab: Atezolizumab 840 mg IV over 60 minutes Day 15 of Cycle 1 then Day 1 and Day 15 of subsequent Cycles
  Radiation: Radiation 8 Gy will be given in 3 fractions QOD beginning Day 12, 13 or 14 of Cycle 1 but 24-72 hours prior to 1st dose of Atezolizumab
Period: Overall Study
Arm/Group | Study Treatment Arm
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Study Treatment Arm
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) by RECIST 1.1
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST): Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Progressive Disease (PD) >= 20% increase in tumor burden relative to nadir or the appearance of one or more new lesions; Stable Disease (SD), not meet criteria for CR/PR/PD.
  ORR is defined as the proportion of all subjects with confirmed PR or CR according to RECIST 1.1, from the start of treatment until disease progression/recurrence
Time Frame: Up to a maximum of 5 months
Measure: Number; unit: Percentage of participants
Arm/Group | Study Treatment Arm
Number analyzed (Participants) | 1
Percentage of participants | 0

2. Secondary Outcome: Assess Adverse Events
Description: The frequency and severity of all treatment related adverse events for the single enrolled subject are reported by CTCAE v5 term and grade.
Time Frame: Up to a maximum of 12 months.
Measure: Number; unit: participants experiencing adverse event
Arm/Group | Study Treatment Arm
Number analyzed (Participants) | 1
participants experiencing adverse event
  LYMPHOCYTE COUNT DECREASED Grade 3 | 1
  NEUTROPHIL COUNT DECREASED Grade 3 | 1
  WHITE BLOOD CELL DECREASED 3 | 1
  ANEMIA Grade 2 | 1
  DIARRHEA Grade 1 | 1
  PLATELET COUNT DECREASED Grade 1 | 1

3. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression free survival (PFS) is defined as the day of study treatment initiation until disease progression by RECIST 1.1 or death whichever occurs first.
Time Frame: Time of treatment start until the criteria for disease progression or death, up to a maximum of 5 months.
Measure: Number; unit: Months
Arm/Group | Study Treatment Arm
Number analyzed (Participants) | 1
Months | 4.4

4. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is defined as the time from treatment start until death or date of last contact.
Time Frame: Time of treatment start until death, up to a maximum of 12 months.
Measure: Number; unit: Months
Arm/Group | Study Treatment Arm
Number analyzed (Participants) | 1
Months | 11.73

5. Secondary Outcome: ORR by Immune-related RECIST (irRECIST)
Description: Per Immune-Related RECIST (irRECIST): Complete Response(irCR), Disappearance of all measurable and non-measurable lesions; Partial Response (irPR) >=30% decrease in tumor burden relative to baseline; Progressive Disease (irPD), >= 20% increase in tumor burden relative to nadir or the appearance of one or more new lesions confirmed by a consecutive assessment at least 4 week after first documentation; Stable Disease (irSD), not meeting criteria for irCR or irPR, in absence of irPD ORR is defined as the proportion of all subjects with CR and PR determined as per irRECIST
Time Frame: Up to a maximum of 5 months
Measure: Number; unit: Percentage of participants
Arm/Group | Study Treatment Arm
Number analyzed (Participants) | 1
Percentage of participants | 0

6. Secondary Outcome: Duration of Overall Response (DOR)
Description: DOR is defined as the time from the measurement criteria are met for complete or partial response (whichever status is recorded first) until the date of recurrent or disease progression.
Time Frame: Up to a maximum of 5 months
Population: No subject achieved CR or PR. Therefore Duration of Response cannot be calculated.
Arm/Group | Study Treatment Arm
Number analyzed (Participants) | 0

7. Secondary Outcome: Disease Control Rate (DCR)
Description: Disease control rate (DCR) is defined as the percentage of patients with advanced or metastatic cancer who have achieved complete response, partial response and stable disease.
Time Frame: Up to a maximum of 5 months
Measure: Number; unit: Percentage of participants
Arm/Group | Study Treatment Arm
Number analyzed (Participants) | 1
Percentage of participants | 100

8. Secondary Outcome: Time to Progression (TTP)
Description: Time to progression (TTP) is defined as the day of study treatment initiation until disease progression by RECIST 1.1.
Time Frame: Up to a maximum of 5 months
Measure: Number; unit: Months
Arm/Group | Study Treatment Arm
Number analyzed (Participants) | 1
Months | 4.4

9. Secondary Outcome: Best Overall Tumor Response
Description: Best overall tumor response is defined as the best response recorded from the start of the study treatment until disease progression/recurrence.
Time Frame: Time of treatment start until the criteria for disease progression, up to a maximum of 5 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Study Treatment Arm
Number analyzed (Participants) | 1
Participants
  PR (Partial Response) | 0
  SD (Stable Disease) | 1
  CR(Complete Response) | 0
  PD (Progressive Disease) | 0

ADVERSE EVENTS:
Time Frame: Up to a maximum of 12 months.
Arm/Group | Study Treatment Arm
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Treatment Arm (N=1)
ANEMIA (Blood and lymphatic system disorders) | 1 (2)
DIARRHEA (Gastrointestinal disorders) | 1 (1)
LYMPHOCYTE COUNT DECREASED (Investigations) | 1 (2)
NEUTROPHIL COUNT DECREASED (Investigations) | 1 (1)
PLATELET COUNT DECREASED (Investigations) | 1 (1)
WHITE BLOOD CELL DECREASED (Investigations) | 1 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-10): https://cdn.clinicaltrials.gov/large-docs/55/NCT04690855/Prot_SAP_000.pdf